CLINICAL TRIAL: NCT04408612
Title: Dyspnea in Stable Patients With Coronary Artery Disease: Causes and Opportunities for Early Differential Diagnosis.
Brief Title: Dyspnea in Stable Patients With Coronary Artery Disease.
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 01-05/20
Record Dates: First submitted 2020-05-10; First posted 2020-05-29 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Dyspnea; Coronary Artery Disease
Keywords: Dyspnea; Stable coronary artery disease; Heart failure; Diastolic stress test
MeSH Terms: conditions — Dyspnea; Coronary Artery Disease; Heart Failure | interventions — Tooth Exfoliation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NT-proBNP, hsTroponin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyspnea in stable coronary artery disease: Stable patients with dyspnea and coronary artery disease
  Interventions: Diagnostic Test: Scales for assessment of symptoms

INTERVENTIONS:
Diagnostic Test: Scales for assessment of symptoms — Medical Research Council Dyspnea scale, the visual analogue scale of dyspnea, Borg scale, modified "dictionary" of dyspnea, G. Rose questionnaire, Seattle Angina Questionnaire, Framingham criteria for chronic heart failure, the SHOCK scale.

SUMMARY:
Single-centre prospective study to characterize causes of dyspnea in stable patients with coronary artery disease and evaluate the possibility to determine the cause of dyspnea before in-depth examination.

DETAILED DESCRIPTION:
Stable patients with dyspnea and coronary artery disease will be included in this single-centre prospective study. In addition to routine clinical examination patients will be interviewed to determine the nature of shortness of breath, angina, presence of chronic heart failure or anxiety using the Medical Research Council Dyspnea scale, the visual analog scale of dyspnea, Borg scale, modified "dictionary" of dyspnea, G. Rose questionnaire, Seattle Angina Questionnaire, Framingham criteria for chronic heart failure and the SHOCK scale. During the subsequent in-depth examination including thyroid hormones, NT-proBNP, hsTroponin, ECG monitoring, six-minute walk test, stress-echo with a diastolic stress test, spirometry and coronary angiography (if necessary) main reason for dyspnea will be established. Possibilities of early (before in-depth examination) determination the reason for dyspnea in stable patients with coronary artery disease will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients with shortness of breath and established diagnosis of coronary artery disease (at least 1 of the following signs):

   * history of myocardial infarction;
   * typical angina without suspected other cause of pain;
   * myocardial ischemia documented by ECG changes during symptoms and/or by results of the stress test;
   * coronary artery stenosis >50% according to coronary angiography.
2. Signed informed consent.

Exclusion Criteria:

1. Acute coronary syndrome (myocardial infarction, unstable angina) in the previous month.
2. Hospitalization with decompensation of CHF in the previous 6 months (including CHF decompensation as the main reason for current hospitalization).
3. Diseases with an unfavourable prognosis (terminal CKD, CHF NYHA IV, a lung disease with severe respiratory failure).
4. Contraindications to bicycle stress echocardiography.
5. Atrial Fibrillation at the time of hospitalization, when the decision not to restore the sinus rhythm.
6. Mental illnesses and disorders, dementia, drug or alcohol dependence.
7. Known oncological diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stable patients with dyspnea and established coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Myocardial ischemia as a reason of dyspnea | up to 1 month
  Number of patient with dyspnea related to myocardial ischemia

SECONDARY OUTCOMES:
Other causes of dyspnea | up to 1 month
  Number of patient with non-ischemic reasons for dyspnea (heart failure, pulmonary disease, arrhythmias, psychogenic, mixed or undetermined cases).
Adverse events | 6 months
  Composite of death, myocardial infarction, stroke and rehospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre for Therapy and Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided